CLINICAL TRIAL: NCT01118039
Title: A Phase II Study Assessing SU-011248 in Previously Untreated Patients With Advanced Urothelial Cancer Ineligible for Cisplatin-Based Chemotherapy
Brief Title: Sunitinib Malate in Treating Patients With Locally Recurrent, Locally Advanced, Unresectable, or Metastatic Urinary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital del Mar (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: HDM-SU-011248; CDR0000671673 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2005-005115-16; PFIZER-HDM-SU-011248
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2012-09

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: localized transitional cell cancer of the renal pelvis and ureter; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent transitional cell cancer of the renal pelvis and ureter; transitional cell carcinoma of the bladder; distal urethral cancer; proximal urethral cancer; recurrent urethral cancer; recurrent bladder cancer; stage IV bladder cancer; stage III bladder cancer; urethral cancer associated with invasive bladder cancer; stage III urethral cancer; stage IV urethral cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Sunitinib; Immunohistochemistry

INTERVENTIONS:
Drug: sunitinib malate
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Sunitinib malate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying the side effects of giving sunitinib malate and to see how well it works in treating patients with locally recurrent, locally advanced, unresectable, or metastatic urinary tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the time to disease progression (defined as the time from diagnosis of metastatic urothelial carcinoma until first confirmed progression of the disease) in patients with locally recurrent, locally advanced, unresectable, or metastatic urothelial cancer treated with sunitinib malate and ineligible for cisplatin-based chemotherapy.
* To determine the safety of this drug in these patients.

Secondary

* To determine the progression-free survival of patients treated with this drug.
* To determine the overall response rate in patients treated with this drug.
* To determine the overall survival of patients treated with this drug.
* To determine the time to treatment failure in patients treated with this drug.
* To determine the pharmacodynamic profile of this drug in pre- and post-treatment serum and tumor tissue (i.e., IL8, VEGF, MMP9, bFGF, p27, Ki-67, and apoptosis [H/E]) at week 6, and if possible, at time of progression.
* To determine the quality of life of patients treated with this drug using the QLQ-C30 version 3 questionnaire.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate once daily on days 1-28. Treatment repeats every 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients complete quality-of-life questionnaire (EORTC QLQ-C30) before, during, and at the end of study treatment.

Serum and tumor tissue samples are collected at baseline and after study treatment for pharmacodynamic studies. Samples are analyzed for markers (i.e., IL8, VEGF, MMP9, bFGF, p27, Ki-67, and apoptosis [H/E]) via immunohistochemistry.

After completion of study treatment, patients are followed for 28 days and then every 2 months for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed transitional cell carcinoma of the urinary tract meeting ≥ 1 of the following criteria:

  * Unresectable, locally recurrent disease

    * Locally recurrent disease must not be amenable to resection or radiotherapy with curative intent
  * Locally advanced or metastatic disease

    * No prior chemotherapy for advanced disease
* Ineligible (unfit) for cisplatin-based chemotherapy due to creatinine clearance < 60 mL/min but > 30 mL/min
* Measurable or nonmeasurable disease according to RECIST criteria

  * Measurable lesions that have been previously irradiated will not be considered target lesions unless increase in size has been observed following completion of radiation therapy

PATIENT CHARACTERISTICS:

* See Disease Characteristics
* ECOG performance status 0-1
* Life expectancy > 12 weeks
* Absolute neutrophil count ≥ 1,500/μL
* Platelet count ≥ 100,000/μL
* Hemoglobin ≥ 9.0 g/dL
* Total serum bilirubin ≤ 1.5 times upper limit of normal (ULN)
* Serum creatinine ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN (≤ 5 times ULN if liver function abnormalities are due to underlying malignancy)
* Serum albumin ≥ 3.0 g/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during study therapy
* No diagnosis of a second malignancy within the past 3 years except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix
* None of the following within the past 12 months:

  * Myocardial infarction
  * Severe/unstable angina
  * Coronary/peripheral artery bypass graft
  * Congestive heart failure
  * Cerebrovascular accident, including transient ischemic attack
  * Pulmonary embolus
* No ongoing cardiac dysrhythmias (NCI CTCAE grade ≥ 2), atrial fibrillation of any grade, or QTc interval > 450 msec (males) or > 470 msec (females)
* No hypertension that cannot be controlled by medications (> 150/100 mm Hg despite optimal medical therapy)
* No known HIV infection
* No other severe acute or chronic medical or psychiatric condition or laboratory abnormality that would impart, in the judgment of the investigator, excess risk associated with study participation or study drug administration, or which would make the patient inappropriate for entry into this study

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all acute toxic effects of prior therapy or surgical procedures to grade ≤ 1 (except alopecia)
* At least 3 weeks since prior major surgery, radiotherapy, or systemic therapy (except palliative radiotherapy to non-target metastatic lesions)
* Not enrolled in a dialysis program or anticipating a need for dialysis
* No prior chemotherapy regimen or biological treatment for locally advanced or metastatic transitional cell carcinoma of the urinary tract
* No prior treatment on another sunitinib malate clinical trial
* No prior tyrosine kinase inhibitors, VEGF inhibitors, or other angiogenic inhibitors
* No prior high-dose chemotherapy requiring hematopoietic stem cell rescue
* No prior radiotherapy to > 25% of the bone marrow
* No concurrent treatment on another clinical trial
* No concurrent treatment with therapeutic doses of acenocoumarol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2006-07; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Time to disease progression
Safety

SECONDARY OUTCOMES:
Progression-free survival
Overall response rate
Overall survival
Time to treatment failure
Pharmacodynamic profile
Quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Bellmunt, MD, PhD — Hospital del Mar
Locations (4):
- Spain (4):
  - Hospital Del Mar, Barcelona
  - Hospital de la Santa Cruz i Sant Pau, Barcelona
  - Hospital Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid